CLINICAL TRIAL: NCT00699868
Title: Cellular Immunity, Cytomegalovirus Infection and Septic Shock in ICU Patients
Brief Title: Immune Response and Cytomegalovirus in Intensive Care Unit (ICU) Patients
Acronym: 2006/25
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Assistance Publique Hopitaux De Marseille, Assistance Publique Hopitaux De Marseille
Model: Parallel | Masking: None
Other Study IDs: 2007-A01197-46
Record Dates: First submitted 2008-06-13; First posted 2008-06-18 (Estimated); Last update posted 2012-06-04 (Estimated); Status verified 2012-06

CONDITIONS: Cytomegalovirus Infection
MeSH Terms: conditions — Cytomegalovirus Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Infection to CMV
  Interventions: Other: Sampling of blood, phenotypic analysis sub-populations NK by cytometric of stream in multiple markings
- 2 (Other): Group "control CMV"
  Interventions: Other: Sampling of blood, phenotypic analysis sub-populations NK by cytometric of stream in multiple markings

INTERVENTIONS:
Other: Sampling of blood, phenotypic analysis sub-populations NK by cytometric of stream in multiple markings — Sampling of blood
  Arms: 1
Other: Sampling of blood, phenotypic analysis sub-populations NK by cytometric of stream in multiple markings — Sampling of blood
  Arms: 2

SUMMARY:
This prospective study evaluate the immune status of patients admitted in ICU.CMV remains dormant in the body, but in people with immune deficiency, CMV could reactivate and cause life-threatening pneumonia.

DETAILED DESCRIPTION:
Candidates will be screened with medical history and blood tests.Then, 2 groups of 20 patients (with or without CMV reactivation) matched for CMV status will be compared for their immune system against CMV.

ELIGIBILITY:
Inclusion Criteria:

* Age more than 18-year-old
* Informed consent

Exclusion Criteria:

* minors,
* pregnant or lactating women,
* adults under guardianship,
* immunosuppression at the entrance to resuscitation,
* AIDS

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2008-03; Primary Completion 2011-01 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Bring to light the quantitative and qualitative immunological modifications of the present cells NK before the arisen of an infection to CMV | 24 months

SECONDARY OUTCOMES:
Bring to light the quantitative and qualitative immunological modifications of cells NK in the consequences of an infectious shock | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Marie FOREL, MD, Principal Investigator — Assistance Publique des Hôpitaux de Marseille
Locations (1):
- Hôpital de Sainte Marguerite- Service de Réanimation Médicale, Marseille, France

REFERENCES:
- [Derived] Matta J, Baratin M, Chiche L, Forel JM, Cognet C, Thomas G, Farnarier C, Piperoglou C, Papazian L, Chaussabel D, Ugolini S, Vely F, Vivier E. Induction of B7-H6, a ligand for the natural killer cell-activating receptor NKp30, in inflammatory conditions. Blood. 2013 Jul 18;122(3):394-404. doi: 10.1182/blood-2013-01-481705. Epub 2013 May 17. PMID 23687088
- [Derived] Forel JM, Chiche L, Thomas G, Mancini J, Farnarier C, Cognet C, Guervilly C, Daumas A, Vely F, Xeridat F, Vivier E, Papazian L. Phenotype and functions of natural killer cells in critically-ill septic patients. PLoS One. 2012;7(12):e50446. doi: 10.1371/journal.pone.0050446. Epub 2012 Dec 6. PMID 23236375